CLINICAL TRIAL: NCT04366609
Title: The Relationship Between CES1 Genotype and Methylphenidate Response in Children With ADHD - INDICES Work Package 6
Status: Completed | Type: Observational
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Copenhagen University Hospital, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: H-B-2009-026
Record Dates: First submitted 2020-03-30; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2012-01

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from saliva collected in the Oragene OG-250 DNA kit (DNA Genotek Inc., ON, Canada).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ADHD patients: Treatment of young ADHD patients with methylphenidate following The Danish guidelines, which are similar to The NICE guidelines: use of an initial low oral dose of MPH and an up-titration period of at least 4 weeks, until no further effect is measured on a standard ADHD rating scale, or the appearance of intolerable ARs, or a maximum dose of 2.1 mg/kg/day.
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate — Treatment with methylphenidate through dose escalation
  Other Names: Medikinet - N06BA04; Motiron - N06BA04

SUMMARY:
This is a prospective observational study of a cohort of children diagnosed with Attention Deficit Hyperactive Disorder (ADHD) and followed with weekly assessments during the first 12 weeks of Methylphenidate (MPH) treatment, and after three years.

The overall aim is to gain knowledge in order to develop guidelines for more individualized treatments with (MPH), obtain a better drug response, and reduce the risk of adverse reactions, in order to improve adherence and long-term outcome.

DETAILED DESCRIPTION:
The study has three aims:

1. Examine the effect of carboxylesterase 1 (CES1) genotype in children with ADHD on the effectiveness and adverse reactions of treatment with MPH.
2. Study predictors for the short- and long-term outcome in childhood ADHD
3. Examine the long-term outcome with respect to ADHD symptoms, and impairment in daily functioning in the cohort

The specific aims are to:

* Describe the treatment response during the first 12 weeks after initiation of IR-MPH treatment, based on weekly clinician- rated ADHD core symptoms, the rate of normalisation/ borderline normalisation of ADHD core symptoms, adverse reactions, daily and social functioning, and measures of sustained attention.
* Describe the three-year outcome, based on parent rated ADHD core- and behavior symptoms, and level of impairment in daily functioning.
* Provide information about predictors for outcome after 12 weeks: clinical characteristics at entry (sex, age group, global severity of psychiatric disorder, psychiatric comorbidity, subtype of ADHD diagnoses), and predictors for outcome after three years: sex, age group, baseline severity of ADHD- and behavior symptoms, IQ, parental psychiatric disorder, maternal educational level, and time to treatment response.
* Determine the end-dose of IR-MPH after 12 weeks of treatment.
* Systematically sequence the CES1 gene and associate the identified genotypes of this gene with treatment responses, including dosage of IR-MPH

ELIGIBILITY:
Inclusion Criteria:

* MPH naïve
* recent ICD-10 diagnosis of hyperkinetic disorder (F90.0-90.9) or attention deficit disorder without hyperactivity (F98.8)
* clinical indication for treatment with IR-MPH

Exclusion Criteria:

* mental retardation (ICD-F70.X or IQ < 70)
* previous treatment with drugs metabolised by carboxylesterase 1 (CES1)
* severe comorbid psychiatric or somatic disease that resulted in contraindication for treatment with MPH
* language barriers
* lack of informed consent.

Specific additional exclusion criteria for genetic analyses:

* Non-caucasian
* Lack of DNA
* Consanguine patients
* Variants with a minor allele frequency (MAF) above 0.05 or not in Hardy-Weinberg equilibrium

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 207 MPH naïve boys and girls aged 7-12 years with a recent ICD-10 diagnosis of hyperkinetic disorder (F90.0-90.9) or attention deficit disorder without hyperactivity (F98.8) and clinical indication for treatment with IR-MPH.
  Patients referred to the Child and Adolescent Mental Health Centre, Mental Health Services (Capital Region of Denmark) in the period from 1st of May 2012 to 1st August 2014, and who were suspected of having ADHD were consecutively screened for study eligibility.
Sampling Method: Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2014-08-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Investigator rated ADHD-RS score | Week 0 to 12
  Psychometric instrument: 18 item clinician rated; Inattention subscale: 9 items, [range 0-27]. Hyperactivity-Impulsivity subscale: 9 items [range 0-27], evaluated on a four-point Likert scale from 0 (none = never or rarely) to 3 (severe = very often). Higher score, worse outcome. Normalisation: T-score<60, Borderline normalisation: T-score 60-70.

SECONDARY OUTCOMES:
Clinical Global Impression Severity scale (CGI-S) | Week 0 and 12
  Psychometric instrument: The clinician-rated CGI-S is a seven-point Likert scale, rated 1 (normal, not ill at all) to 7 (among the most extremely ill patients)A beneficial symptom reduction was defined by a CGI-S score of 1 or 2 (normal, not ill at all or borderline ill).
Clinical Global Impression Improvement (CGI-I) | Week 4-8-12
  Psychometric instrument, clinician-rated CGI-I seven-point Likert scale rated from 1 (very much improved) to 7 (very much worse). A beneficial symptom reduction was defined by a CGI-I score of 1 or 2 (very
Test of Variables of Attention (TOVA) | Week 0 and 12
  Computerized, continuous performance test, number of commission errors (response to non-target), number of omission errors (non-response to target), the response time in microseconds, and the variability of response time in correct responses to target were measured over the 21.6-minute-long test used as total raw scores.
Parent rated ADHD-RS | Week 0-4-8-12, year 3
  Psychometric instrument: Inattention subscale: 9 items, [range 0-27]. Hyperactivity-Impulsivity subscale: 9 items [range 0-27]. Conduct problems subscale: 8 items, [range 0-24]. Higher score, worse outcome.
Teacher rated ADHD-RS | Week 0-4-8-12
  Psychometric instrument: Inattention subscale: 9 items, [range 0-27]. Hyperactivity-Impulsivity subscale: 9 items [range 0-27]. Conduct problems subscale: 8 items, [range 0-24]. Higher score, worse outcome.

OTHER OUTCOMES:
Weiss Functional Impairment Rating Scale - Parent version (WFIRS-P). | Week 0 and 12, year 3
  Psychometric instrument: WFIRS-P is a parent-rated questionnaire, with 50 questions about a child's daily and social functioning in six different domains of a child's life: family (10 items), learning and school (10 items), activities of daily living (10 items), self-concept (3 items), social activities (7 items), and risky activities (10 items). It is evaluated on a four-point Likert scale from 0 (never or not at all) to 3 (very often or very much). Single item scores = 2-3 signal impairment (> 2 SD). Higher score, worse outcome.
Barkley's Stimulant Side Effect Rating Scale (BSSERS-C) | Week 0 to 12
  Psychometric instrument: 17 effect items rated by the clinician, based on information from patients, parents, and clinical observations: insomnia, nightmares, staring, talks less, disinterested in others, reduced appetite, irritable, stomachaches, headaches, drowsiness, sadness, prone to crying, anxious, nail biting, euphoria, dizziness, and tics/nervous movements. BSSERS-C is a 10-point Likert scale rated from 0 (problem absent) to 9 (problem evokes serious impairment). Severities of ARs were calculated as the sum of problem scores on the 17-item BSSERS-C. Significant changes in single items were also explored (e.g., reduced appetite; 1 item, range 0-9).
Child Behaviour Check List (CBCL) | Week 0
  Psychometric instrument: Parent rated. Externalizing score: 35 items [range 0-70]. Internalizing score: 32 items [range 0-64]. Total problem score: 118 [range 0-236].
Teacher Report Form (TRF) | Week 0
  Psychometric instrument: Teacher rated. Externalizing score, 34 items [range 0-68]. Internalizing score: 34 items [range 0-68]. Total problem score: 118 [range 0-236].
MPH dose required for "Borderline normalisation" on ADHD-RS | Week 0 to 12
  The IR-MPH doses were individually titrated, based on the weekly evaluations of symptom reductions and ARs (and the body weight of a child), which were carried out by the clinical investigator. The dose of IR-MPH (mg/kg/day) at the end of the study was registered. Dose required for T-score of 60-70 on ADHD-DSM-IV-RS.
MPH dose required for normalisation on ADHD-RS | Week 0 to 12
  The IR-MPH doses were individually titrated, based on the weekly evaluations of symptom reductions and ARs (and the body weight of a child), which were carried out by the clinical investigator. The dose of IR-MPH (mg/kg/day) at the end of the study was registered. Dose required for T-score < 60 on ADHD-DSM-IV-RS.
Genetic analyses | Week 0
  The genetic analyses of CES1 were carried out using PCR and sequencing.
Body weight | Week 0-4-8-12
  Body weight in kilograms
Height | Week 0-4-8-12
  Height in centimeters
Heart rate | Week 0-4-8-12
  Heart rate, bp/m
Blood pressure | Week 0-4-8-12
  Both diastolic blood pressure, mmHg, and Systolic blood pressure, mmHg, measured after 10 minutes of rest with a sphygmomanometer (nonelectrical) three times and the average of the last two measures is used
Reduced appetite: single item, [range 0-9]. | Week 0-4-8-12
  Single item of psychometric instrument Barkley's Stimulant Side Effect Rating Scale (BSSERS-C), [range 0-9]. Higher value, worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Pia Jeppesen, PhD, MD, Principal Investigator — Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital; Tine B Houmann, MD, Study Director — Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Houmann TB, Kaalund-Brok K, Clemmensen L, Petersen MA, Plessen KJ, Bilenberg N, Verhulst F, Jeppesen P; INDICES. Early treatment response as predictor of long-term outcome in a clinical cohort of children with ADHD. Eur Child Adolesc Psychiatry. 2024 Feb;33(2):357-367. doi: 10.1007/s00787-023-02158-z. Epub 2023 Feb 16. PMID 36795232
- [Derived] Kaalund-Brok K, Houmann TB, Hebsgaard MB, Lauritsen MG, Lundstrom LH, Gronning H, Darling L, Reinert-Petersen S, Petersen MA, Jepsen JRM, Pagsberg AK, Plessen KJ, Rasmussen HB, Jeppesen P; INDICES. Outcomes of a 12-week ecologically valid observational study of first treatment with methylphenidate in a representative clinical sample of drug naive children with ADHD. PLoS One. 2021 Oct 21;16(10):e0253727. doi: 10.1371/journal.pone.0253727. eCollection 2021. PMID 34673771

DOCUMENTS (1):
  • Study Protocol (2012-03-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT04366609/Prot_000.pdf